CLINICAL TRIAL: NCT06762041
Title: A Cohort Study to Elucidate the Effects of Metformin on Androgens and Other Steroid Hormones in Affected Subjects With Autism - a First Pilot Study
Brief Title: Effects of Metformin on Androgens and Other Steroid Hormones in Affected Subjects With Autism
Acronym: Metformin
Status: Not yet recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: Steroidlabs; Lindenhofhospital Berne (Other: Lindenhofhospital Berne)
Record Dates: First submitted 2024-11-21; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Steroid hormone concentrations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Metformin Treatment
  Interventions: Drug: Metformin treatment

INTERVENTIONS:
Drug: Metformin treatment — Interested subjects with autism are treated with metformin with a standard dosage
  Other Names: Metformin treatment in subjects with autism

SUMMARY:
Autism is diagnosed with increasing frequency in recent years despite remaining uncertainty concerning the cause. The disorder is characterized by deficits in social behavior, a lack of communication skills, and repetitive and stereotypical interests. As part of the research, It attempted to pursue the hypothesis that the disorder is signed by an endocrine involvement. Therefore, the original description of Hans Asperger was analyzed first. This was followed by comprehensive steroid hormone analyses in girls and boys with autism. Based on the assumption that steroid hormones are involved, dysregulation of the adrenal gland for all metabolite classes - mineralocorticoid, glucocorticoid, androgen - were identified. The subsequently followed animal experiments yielded to the conclusion that a dysregulation of the hypothalamic-pituitary system might be responsible for the autistic behavior. This is also probably associated with overactivity of 17/20 lyase, an orchestrating enzyme of oxidative stress, which is driven by p38. It is suspected that the increased oxidative stress is of mitochondrial origin and thus other metabolic cascades are involved. Due to the developed understanding of the suspected dysregulation, new therapeutic options for treatment are opening up, with metformin in particular - known for its antiandrogenic effect used in poly cystic ovarian syndrome - appearing to have the best effect on social withdrawal in the developed mouse model. Initial urine analyses allow the assumption that metformin directly influences steroidogenesis, and thus opens up the possibility of a clinical trial for affected subjects with autism.

DETAILED DESCRIPTION:
To date, the etiopathogenesis or the biochemical basis of social withdrawal behavior have not been conclusively clarified and accordingly the treatment options are not exhausted. Investigators know from analyzes of those affected by the most severe form of social impairment respectively from subjects with autism that there appears to be a change in the cholesterol-dependent steroid metabolism. Furthermore, it can be assumed that treatment with different substances could be promising. Metformin seems to cause a direct inhibition of the androgen synthesis pathways while parallel influencing social behavior. In principle, Metformin is mainly used to treat Diabetes mellitus type 2. It is a biguanide drug that has been used for more than 60 years. Studies have shown that metformin improves mortality rates in diabetes patients, and younger studies show additional effects in treating cancer, obesity, nonalcoholic fatty liver disease, polycystic ovary syndrome and metabolic syndrome.Treatment with metformin mimics some of the benefits of caloric restriction, such as improved physical performance while yielding to increased insulin sensitivity and reduced low-density lipoprotein and cholesterol levels. Furthermore, as chronic inflammation is also influenced by exercise training it is allowed to assume similar mechanism of Metformin and physical activity. At a molecular level, metformin increases activated protein kinase activity and increases antioxidant protection, resulting in reductions in both oxidative damage accumulation and chronic inflammation thereby mimicking positive effects of endurance training.In consequence, it was indicated that these actions may contribute to the beneficial effects of metformin on health- and lifespan. Focusing on neurologic diseases affected by Metformin positive effects on Alzheimer's disease were shown. Metformin attenuated spatial memory deficit, neuron loss in the hippocampus and enhanced neurogenesis in mice. In another mouse model the metformin treatment counteracted the development of depression-like behaviors in mice suffering social defeat stress when administered. This directly yields to the aim of the study: to assess effects of Metformin on steroid hormones in subjects affected with autism.

ELIGIBILITY:
The inclusion criteria:

* Diagnosis with autism according to DSM-V.
* Written informed consent

The exclusion criteria:

* Clinically significant concomitant disease states (e.g. advanced renal failure, hepatic Dysfunction - risk factor of lactate acidosis)
* Significant musculoskeletal disease
* Active infection
* Immunosuppressive medical therapy
* Known or suspected non-compliance, drug or alcohol abuse
* Pregnant or breastfeeding mothers are excluded
* Inability to follow the procedures of the study, e.g. due to insufficient language skills, psychological disorders, very severe dementia inability to report adequately

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with autism
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Steroid hormone concentrations of total androgens | After 6-9 month of treatment with Metformin
  Steroid hormones

CONTACTS AND LOCATIONS:
Overall Officials: Markus Mohaupt, Prof. Dr., Study Director — University of Berne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gasser BA, Kurz J, Dick B, Mohaupt MG. Steroid Metabolites Support Evidence of Autism as a Spectrum. Behav Sci (Basel). 2019 May 9;9(5):52. doi: 10.3390/bs9050052. PMID 31075898
- [Background] Gasser BA, Kurz J, Senn W, Escher G, Mohaupt MG. Stress-induced alterations of social behavior are reversible by antagonism of steroid hormones in C57/BL6 mice. Naunyn Schmiedebergs Arch Pharmacol. 2021 Jan;394(1):127-135. doi: 10.1007/s00210-020-01970-7. Epub 2020 Sep 7. PMID 32894324
- [Background] Gasser B, Escher G, Calin AE, Deppeler M, Marchon M, Kurz J, Mohaupt M. Are steroid hormones and autistic traits affected by metformin? First insights from a pilot. Compr Psychoneuroendocrinol. 2023 Jul 29;16:100196. doi: 10.1016/j.cpnec.2023.100196. eCollection 2023 Nov. PMID 37577184
- [Background] Gasser B, Escher G, Calin AE, Deppeler M, Marchon M, Mistry HD, Kurz J, Mohaupt MG. Prior to versus after Metformin Treatment-Effects on Steroid Enzymatic Activities. Life (Basel). 2023 Apr 27;13(5):1094. doi: 10.3390/life13051094. PMID 37240739